CLINICAL TRIAL: NCT06636812
Title: The Effects of Single-dose Losartan on the Processing of Emotional Information in Healthy Adolescents: a Randomised Controlled Study
Brief Title: Losartan and Emotional Processing in Young People
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford Health Biomedical Research Centre (OH BRC) support scheme (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R79545
Record Dates: First submitted 2024-09-23; First posted 2024-10-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-09

CONDITIONS: Emotional Processing
Keywords: emotional processing; anxiety; adolescents
MeSH Terms: conditions — Anxiety Disorders | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Parallel randomised experimental medicine trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- losartan (Experimental): single-dose losartan potassium (Cozaar; weight-adjusted 25mg or 50mg)
  Interventions: Drug: Losartan potassium
- Placebo (Placebo Comparator): Microcellulose placebo in identical capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan potassium — Single dose losartan (25mg or 50 mg, weight-adjusted), encapsulated identically to placebo
  Arms: losartan
Other: Placebo — Single tablet encapsulated identically to placebo
  Arms: Placebo

SUMMARY:
This study explores the effects of single-dose losartan (50mg) versus placebo on emotional processing in young healthy volunteers.

DETAILED DESCRIPTION:
Compared to children and adults, adolescents are most likely to develop an anxiety disorder and less likely to respond to even the most effective treatment - exposure therapy. Similarly, fear extinction - the laboratory equivalent to exposure therapy - is impaired in this young age group. Animal and human research suggests that such deficits in fear reduction may be underpinned by insufficient functioning of the ventromedial prefrontal cortex (vmPFC) during adolescence as part of normative development.

A single dose of losartan, a commonly prescribed blood pressure drug targeting the renin-angiotensin system, has been shown to enhance fear extinction in adult humans (Zhou et al. 2019). Most importantly, such effects are seen to be driven by improved vmPFC function following losartan (Zhou et al. 2019). Our own work in adults has also demonstrated rapid beneficial effects of single-dose losartan on other neurocognitive markers relevant to anxiety and treatment response, while not revealing any adverse reactions (Reinecke et al., 2018; Pulcu et al., 2019; Shkreli et al., 2020). These findings suggest that the renin-angiotensin system plays a key role in the extinction of anxiety, and that adding losartan to exposure therapy for anxiety in humans might have synergistic effects.

In this double-blind, randomized between-group study, we will investigate the effects of a single dose of losartan (weight-adjusted: 50mg if over/ 25mg if below 50kg) versus placebo on emotional processing in N=60 healthy volunteers aged 16-20 years. One hour later, when drug-peak plasma levels are reached, participants will work on a battery of computerized tasks, including a fear extinction task and other tasks exploring attention for and learning from neutral and emotional stimuli of differing valence. Results from this study will help us understand how the renin-angiotensin system affects emotional processing in human adolescents, and they will help us identify potential synergistic overlaps with the cognitive mechanisms of effective exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent (for 16 and 17 year olds: assent and parental/ legal guardian consent)
* Non- or light-smoker (< 5 cigarettes a day)
* Ability to attend appointments in Oxford with reasonable travel costs
* Ability/ willingness to provide GP contact details

Exclusion Criteria:

* Past or present DSM-5 axis-I diagnosis (based on SCID results at screening), especially severe psychiatric illness or alcohol or substance dependence
* First-degree family member with severe psychiatric illness
* CNS-medication last 6 weeks (including as part of another study)
* Current blood pressure or other heart medication (especially aliskiren or beta blockers)
* Diagnosis of intravascular fluid depletion or dehydration
* Impaired kidney function (based on blood test at screening, cut-off 75 ml/min/1.73 m2)
* Significant hyperkalaemia (level>=6mEq/L in the absence of sample haemolysis will be considered significant hyperkalaemia)
* Very low blood pressure (defined as repeated (at least three consecutive measurements) measures of blood pressure under standardised conditions where either the systolic or the diastolic blood pressure or both are below 90/50 mmHg (in accordance with established standard definitions: DOI 10.1186/s12887-016-0633-7))
* Body weight below 35kg (as the lower dose of 25mg of losartan only indicated from 35kg)
* Lifetime history of epilepsy or other neurological disease (e.g. ADHD, autism)
* Lifetime history of angioedema, renal artery stenosis, valvular heart disease, recurrent postural/ orthostatic hypotension
* Lifetime history ofsystemic infection, or clinically significant hepatic, cardiac, obstructive respiratory, renal, cerebrovascular, metabolic, endocrine or pulmonary disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Significant loss of hearing that is not corrected with a hearing device Insufficient written and/or spoken English skills
* Women: pregnancy, breast-feeding

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fear Extinction | 1 hour after capsule intake
  fear extinction score, computed as a 5-point Likert scale valence rating (1=unpleasant-5=pleasant) of the CS+ stimulus at the end of extinction minus at the end of acquisition, with larger scores indicating better fear extinction

SECONDARY OUTCOMES:
Pattern Separation | 1 hour after capsule intake
  Lure discrimination index (LDI), calculated as the rate of 'similar' responses to lures minus 'similar' responses to foils, with higher scores indicating better mnemonic discrimination
Cognitive Flexibility | 1 hour after capsule intake
  switch cost, calculated by rank-ordering the differences between each switch trial RT and each participants average RT for all non-switch trials from 1 - 10 (with better and worse bins having values closer to 1 and 10, respectively), and then summing the bin values to compute a total bin score for each participant. Inaccurate responses are penalized by being assigned a score of 20. Smaller bin scores indicate greater accuracy and lower RT.
Reinforcement Learning | 1 hour after capsule intake
  reinforcement learning, calculated as the learning rate from aversive and appetitive decision outcomes. Larger scores indicate better learning from an outcome.
Faces Dot Probe Task | 1 hour after capsule intake
  extradecisional threat bias, calculated by subtracting the extradecisional time parameter for congruent trials from the extradecisional time parameter for incongruent trials. Larger scores indicate a greater degree of vigilance to threat.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Reinecke, PhD, Principal Investigator — University of Oxford
Locations (1):
- Warneford Hospital, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided